CLINICAL TRIAL: NCT04033588
Title: A Prospective, Multi-centre, Non-comparative, Post-market Clinical Follow-up Study to Evaluate the Survivorship, Safety and Performance of the Freedom® Total Knee System in United Kingdom.
Brief Title: Freedom® Total Knee System for Treatment of Osteoarthritis, Rheumatoid Arthritis or Post-traumatic Arthritis
Acronym: Freedom®450
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLSIPL/ Freedom® 450
Record Dates: First submitted 2019-01-23; First posted 2019-07-26 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Knee Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: A prospective, multi-centre, non-comparative, post-market clinical follow-up study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Freedom® Total Knee System (Other): A prospective, multi-centre, non-comparative, post-market clinical follow-up study to evaluate the survivorship, safety and performance of the Freedom® Total Knee System in United Kingdom
  Interventions: Device: Freedom® Total Knee System

INTERVENTIONS:
Device: Freedom® Total Knee System — To evaluate the survivorship, safety and performance of the Freedom® Total Knee System in the treatment of subjects who in the surgeon's opinion require a primary total knee replacement due to severe knee joint pain and loss of mobility due to osteoarthritis, rheumatoid arthritis or post-traumatic arthritis.

SUMMARY:
A prospective, multi-centre, non-comparative, post-market clinical follow-up study to evaluate the survivorship, safety and performance of the Freedom® Total Knee System in the treatment of approximately 450 subjects who in the surgeon's opinion require a primary total knee replacement due to severe knee joint pain and loss of mobility due to osteoarthritis, rheumatoid arthritis or post-traumatic arthritis at upto 15 centers in the United Kingdom (UK). The primary objective of this study is to obtain implant survivorship and clinical outcomes data for commercially available Freedom® Total Knee System used in total knee replacement. Subjects must meet all the study inclusion / exclusion criteria before enrolment in the study. Subjects will be requested to attend out-patients clinic for clinical follow-up (CFU) or approached for telephonic follow-up (TFU) post-operatively as mentioned below.

Clinical & Telephonic Follow-up details:

* 6-8 weeks ± 1week (Clinical follow-up)
* 1 year ± 1 month (Clinical follow-up)
* 3 years ± 6 months (Clinical follow-up)
* 5 years ± 6 month (Clinical follow-up (optional) / Telephonic follow-up)
* 10 years± 6 month (Clinical follow-up (optional) / Telephonic follow-up)

DETAILED DESCRIPTION:
At all the clinical/telephonic follow-up visits i.e. at 8 weeks ± 1week, 1 year ± 1 month, 3 years ± 6 months, 5 years ± 6 months and 10 years ± 6 months implant survivorship and vital signs such as weight, heart rate etc including blood pressure will be recorded. Physical examination, lab measurements (optional), Radiographic assessment, concomitant medication/surgery and AE/SAE should be recorded. Also at all clinical follow ups OKS, KSS, range of motion will be recorded. The post-operative radiographic evaluations will be conducted at 0-8 weeks ± 1 week (which is considered as standard of care), 1 year ± 1 month, 3 years ± 6 months and optionally at 5 years ± 6 months, 10 years ± 6 months and Unscheduled visits, if required. The unscheduled visit is expected in some patients based on the fact that such patients might prone to complications like surgical site infections, venous thrombotic events, acute blood loss causing anaemia, nerve injury, and pain unresponsive to oral analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 years and 75 years.
* Subjects who require unilateral knee prosthesis and have been evaluated as appropriate candidates for a total knee replacement by the investigator.
* Subjects suffering from severe knee joint pain and loss of mobility due to rheumatoid arthritis, osteoarthritis or post-traumatic osteoarthritis.
* Subjects, who in the opinion of the investigator are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow ups.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this clinical investigation.
* Subjects who are known drug or alcohol abuse or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subject with a known sensitivity to device materials.
* Subjects with other significant disabling problems from the muscular-skeletal system other than in the knees (i.e muscular dystrophy, polio, neuropathic joints).
* Subjects with a BMI of 40 or above.
* Subjects with a current or active history of malignancy, active or suspected infection, Paget's disease, renal osteodystrophy, immunologically suppressed or have any other significant medical illness judged by investigator to exclude from study.
* Subject with neuromuscular or neurosensory deficiency that may limit ability of the patient to evaluate the safety and efficacy of the device.
* Female subjects who are pregnant or lactating.
* Subjects who have previously undergone total or unicondylar knee replacement, high tibial osteotomy, ligament reconstruction, open reduction internal fixation (ORIF) or with previous fracture in the ipsilateral knee joint.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 450 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship Kaplan-Meier estimates of survivorship for all components | At 3 years
  Implant survivor-ship will be established by using revision surgery on the operated knee as implant failure.

SECONDARY OUTCOMES:
Oxford Knee Score which consists of 12 questions | At 1 year and 3 years
  Oxford Knee Score is a patient-reported validated outcome measure scoring from 0 - 48. It consists of 12 questions related to patient's own perception of pain and function in the knee being evaluated. Higher the score better the functioning of the knee.
Range of Motion using a standard goniometer | At 1 year and 3 years
  Range of motion will be assessed using a standard goniometer. It will measure the angle between maximum extension and maximum flexion that a patient can achieve in the operated knee.
Knee Society Score | At 1 year and 3 years
  This score consists of points given for pain, range of motion, and stability. It Consists of points given for the ability to walk on level surfaces, and the ability to ascend and descend stairs.Score range of the KSS is from 0 to 100 points for each portion, with higher scores indicating better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Hemant Pandit, FRCS (Orth), Principal Investigator — Chapel Allerton Hospital and University of Leeds

IPD SHARING:
Plan to Share IPD: No